CLINICAL TRIAL: NCT06782815
Title: Study on the Curative Effect and Autonomic Nerve Function of Primary Insomnia Patients with Liver Depression and Spleen Deficiency Type Based on Acupoint Selection of Meridian Theory
Brief Title: Acupoint Selection Based on Meridian Theory in Primary Insomnia of Liver Depression and Spleen Deficiency Type
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuanlong Zhou (Other)
Responsible Party: Sponsor-Investigator, Chuanlong Zhou, Deputy Chief Chinese Physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024ZL531-primary insomnia
Record Dates: First submitted 2024-12-16; First posted 2025-01-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Primary Insomnia
Keywords: Liver stagnation and spleen deficiency type insomnia; Acupuncture; Randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): This group will include 48 patients. Conventional acupuncture, patients take the supine position
  Interventions: Device: Acupuncture
- Acupuncture group (Experimental): This group will include 48 patients. The patient was placed in a supine position.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — acupuncture Baihui, Sishencong ; acupuncture bilateral Qimen, Zhangmen, Hegu, Taichong, reinforcing and reducing, until the acid swelling is obvious,stopped ferforming acupuncture, the needle was retained for 30 min.
  Arms: Control group
Device: Acupuncture — （1）Acupuncture bilateral Tianrong points, obliquely 45 ± 5 ° backward, 1-1.5 inch deep, reinforcing and reducing horizontally, and stop the needle when the auricle has a heat sensation ; （2）Acupuncture at bilateral Tianyou points, pointing to the tip of the nose, with a depth of 0.5-1 inches, flat reinforcing and reducing, until the sense of soreness and distension obviously stops, and the needle is retained for 30 minutes.
  Arms: Acupuncture group

SUMMARY:
The classical literature combined with modern medicine to select acupoints, in order to intervene in the autonomic nerve function of the superior cervical sympathetic ganglion as an opportunity, put forward the meridian acupoints mainly to reconcile the head orifices Ying Wei, acupuncture treatment of primary insomnia clinical research. Heart rate variability ( HRV ), Pittsburgh sleep quality index ( PSQI ), polysomnography ( PSG ) and the MOS item short from health survey ( SF-36 ) were observed. Insomnia Severity Index ( ISI ), Dysfunctional Beliefs and Attitudes about Sleep Scale 16 ( DBAS-16 ), GABA, Glx and other secondary indicators were used to clarify the clinical short-term and long-term efficacy of different acupoints in the treatment of patients with primary insomnia and the intervention effect on HRV.

DETAILED DESCRIPTION:
In this randomized controlled trial, 96 patients with insomnia of liver depression and spleen deficiency type were selected from the Third Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine. All patients will be randomly assigned to the control group or the acupuncture group.

MAIN OUTCOME MEASURES : Pittsburgh Sleep Quality Index ( PSQI ) was used to measure sleep quality, and 36-Item Short Form Health Survey ( SF-36 ) was used to measure quality of life. Secondary outcomes included the Insomnia Severity Index ( ISI ), Sleep Dysfunction Beliefs and Attitudes Scale 16, DBAS-16, GABA and Glx.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnostic criteria of insomnia of liver depression and spleen deficiency type in traditional Chinese medicine :
* In line with the Western diagnostic criteria for insomnia ;
* 18 ≤ age ≤ 40 years old, male or female ;
* patients with a course of more than two weeks ; Note: The above criteria must be met for inclusion in this study.

Exclusion Criteria:

* Insomnia caused by a variety of organic diseases, neurological or psychiatric disorders
* Pregnancy, lactation or drug allergy
* There are more serious primary diseases such as cardiovascular and cerebrovascular diseases, gastrointestinal diseases, endocrine system diseases, or psychiatric patients.
* Patients with coagulation dysfunction and bleeding tendency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep quality measured by Pittsburgh sleep quality index ( PSQI) | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  The patients will be assessed by PSQI Chinese fixed questionnaire at each observation point and the clinical efficacy will be observed.It consists of 19 self-evaluation and 5 other-evaluation items. Only 19 self-evaluation questions are scored, and 19 self-evaluation questions are composed of 7 factors, each factor consists of 7 factors of 0-3 points. '0 ' refers to no difficulty, ' 3 ' refers to very difficult. The total score of ' 21 ' refers to very difficult in all respects. The sum of all factor scores constitutes the total score of the 0-21 scale. The reference boundary value of adult sleep quality problems in China : poor sleep quality : PSQI ≥ 8 ; good sleep quality : PSQI ≤ 7 ; the higher the score, the worse the sleep quality.
Quality of life measure by 36-item short form health survey（SF-36） | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  The patients will be evaluated by SF-36 scale at each observation point. The SF-36 scale is a general scale developed by the American Medical Research Group to evaluate the quality of life. It is widely recognized and widely used in the world. This scale has eight dimensions to evaluate health-related quality of life ( HRQOL ), which belong to two categories of physical health and mental health, namely physiological function ( PF ), role physical ( RP ), bodily pain ( BP ), general health ( CH ), vitality ( VT ), social function ( SF ), role emotional ( RE ), mental health ( MH ). In addition, the SF-36 scale also includes another indicator - health change ( HT ), which is used to evaluate health changes over the past year.Add the scores of each item to the actual score, and then calculate the final score RP according to the following formula. The higher the RP score, the better the health status.

SECONDARY OUTCOMES:
Insomnia Severity Index（ISI） | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  The patients were evaluated by ISI scale at each observation point. According to the total score, the degree of insomnia is divided into the following degrees：The total score between 0 and 7 indicates no clinically significant insomnia, the total score between 8 and 14 indicates subthreshold insomnia, the total score between 15 and 21 indicates clinical insomnia ( moderate to severe ), and the total score between 22 and 28 indicates clinical insomnia ( severe ).
Dysfunctional Beliefs and Attitudes about Sleep Scale 16，DBAS-16 (DBAS-16) | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  There were 16 items in DBAS-16, including 4 factors : an estimated factor for the consequences of insomnia ; worry about sleep factor ; expectation factors of sleep ; cognition factors of insomnia drugs.The lower the total score, the more likely it is that the subjects ' cognition of sleep is biased.
GABA | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  GABA is the most important inhibitory neurotransmitter in the central nervous system. In clinical studies, proton magnetic resonance spectroscopy showed that GABA in the brain of patients with primary insomnia was 30 % lower than that of normal people, and sleep time was prolonged with the increase of GABA content.
Glx | Before treatment, 4 weeks of treatment, and 4 weeks after the end of treatment, three time points were observed.
  Glutamate glutamine complex ( Glx ) is glutamic acid ( Glu ) + glutamine ( Gln ). Glu is the main excitatory neurotransmitter, maintaining the excitability of organisms. In the clinical study, the content of Glu in the brain of insomnia patients was analyzed by EEG ultra-slow fluctuation technique. The results showed that the content of Glu in insomnia patients increased.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No